CLINICAL TRIAL: NCT00766051
Title: The Efficacy of Neurophysiologically Based Occupational Therapy Intervention in the Neonatal Intensive Care Unit: An Exploratory Study
Brief Title: A Study of Neurophysiologically Based Occupational Therapy Intervention (NBOTI) for Feeding in the NCCU.
Acronym: NBOTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Walden University (Other); Primary Children's Hospital (Other); Mesa State College: Grand Junction, Colorado (Unknown); Politecnico di Milano: P.zza Leonardo da Vinci, 32, 20133 Milano, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23739
Record Dates: First submitted 2008-09-03; First posted 2008-10-03 (Estimated); Results first posted 2012-09-11 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Cerebral Palsy; Sensorimotor Deficits; Sensory Processing Disorder; Feeding Problems; Developmental Coordination Disorder; Picky Eaters; NICU
Keywords: Neurophysiologically Based Occupational Therapy Intervention (NBOTI); NBOTI; NICU; NCCU; Developmental Biology; Critical Period; Brain Development; Sensory Integration; Neurodevelopment; Sensitive Period
MeSH Terms: conditions — Cerebral Palsy; Motor Skills Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): The infants in the intervention group were problem eaters with various diagnosis
  Interventions: Other: The intervention group: Neurophysiologically Based Occupational Therapy Intervention (NBOTI)
- Matched Historical Comparison Group (No Intervention): The matched historical comparison group were also problem eaters and these infants did not receive the neurophysiologically based occupational therapy Intervention.

INTERVENTIONS:
Other: The intervention group: Neurophysiologically Based Occupational Therapy Intervention (NBOTI) — This study included a pre-feeding, feeding, and postural-respiratory protocol, given per the attending physician's order. The interventions were given daily when possible, and the infants FiO2 and heart rate, along with stress behaviors, were monitored prior to, during, and after the NBOTI. The intervention included parent education for feeding, handling, and interaction with their infant, along with nursing training during the feeding session. The occupational therapy investigator partnered with the parents and when the parents were not available, she partnered with the nursing staff.
  Arms: Intervention Group

SUMMARY:
Many critically ill newborns in the neonatal intensive care (NICU) or critical care unit (NCCU) environment develop feeding and movement problems. The purpose of this study was to determine the extent to which neurophysiologically based occupational therapy intervention (NBOTI) for NCCU infants would affect the intervention group's oral feeding and other covariates, such as heart rate variability (HRV) during feeding. The biopsychosocial model provided the study's conceptual framework. The key research question explored whether NBOTI in the NCCU promoted healthy infant development through feeding, movement organization, and parent self-efficacy. This exploratory study with 10 NCCU infants and 10 historical matched controls utilized a mixed method design of qualitatively coded video analysis and inferential statistics such as the t test, the binomial test, hierarchal linear modeling (HLM), and multivariate analysis. Significant differences were obtained between the intervention and comparison groups in the number of days from all tube to all oral feeding before discharge and speed at which the infants gained weight. Longitudinal analyses of the intervention group data were employed to reveal significant trends and pre/post differences in the HRV data along with how quickly the infants ate, parent perceptions of self efficacy and decreased stress in the NCCU. Finally, qualitative findings obtained from videotape analysis provide further evidence that NBOTI was effective in facilitating feeding and promoting development. The recommendations are to replicate this study to validate and expand the findings of the current study. The model for infant care suggested by the findings could contribute to positive social change by fostering positive physical and emotional child development and healthy child-parent and family-caregiver relationships.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common physical disability in childhood (Surveillance of Cerebral Palsy in Europe [SCPE], 2000, 2002; Winter, Autry, Boyle, & Yeargin-Allsopp, 2002),and epidemiological studies of industrialized countries indicate that CP occurs in 2.0 to 2.5 per 1000 live births (Hagberg, Hagberg, Beckung, & Uvebrant, 2001; Paneth & Kiely, 1984; Parkes, Dolk, Hill, & Pattenden, 2001). CP is defined as a movement impairment ranging from mild to severe (Bax et al., 2005; Bobath, 1954; Nelson, 2001); and occurs through social, physical and environmental causal pathways that result in a brain lesion sometime during the ante, peri or post natal period of birth (Stanley, Blair, & Alberman, 2000).

Preterm birth accounts for 40% of all cases of cerebral palsy (Stanley et al., 2000). An infant is born preterm if the birth occurs between 17-36 weeks from their date of conception. Per 1,000 births in the United States between 1989 and 1996, the rate of preterm births increased by 4%, with African American preterm births nearly twice that of whites (Morbidity and Mortality Weekly Report [MMWR], 1999). The rate of preterm birth in the United States is about 10% of all births. Early born preterm infants need organ support in neonatal intensive care unit (NICU) nurseries. Problems encountered by this population due to their undeveloped systems consist of respiratory, cardiac, central nervous system (CNS) vulnerability for damage, feeding and gastrointestinal, and kidney problems (Goldenring, 2004). Very and extremely preterm infants (less than 32 weeks) have the highest rate of developmental disability. Norm referenced cognitive, social, and neuro-developmental test scores at 6 years of age indicated that 80% of extremely preterm infants exhibited mild, moderate, and severe sensorimotor (perceptual-cognitive-motor) disability; with 12% of these infants diagnosed with disabling CP (Marlow, Wolke, Bracewell, & Samara, 2005). Rose, Feldman, & Jankowski, (2002) found that very preterm children needed 30% more time to process visual and somatosensory perceptual information needed for intellectual tasks at 5, 7, and 12 months of age. These discrepancies in efficient processing of sensorimotor stimulation continue into childhood (DeMaio-Feldman, 1994; Feder, et al. 2005) as measured from a child's cognitive responses to their environment (Barlow & Lewandowski, 2000), and internally from mechanisms that provide a foundation for equilibrium and perception such as information generated from within joints, muscles, and skin as tactile-kinesthetic information (Bracewell & Marlow,2002; de Groot, van Hoek, Hopkins, & Touwen, 1993), and as auditory, vestibular, and visual postural-spatial processing (de Graaf, Samsom, Pettersen, Schaaf, van Schie, & de Groot, 2004; De Vries, & De Groot, 2002). In addition to factors such as low birth weight that predispose infants to central nervous system insult (40%), the remaining 60% of infants who are diagnosed with CP suffer from acute insult to the CNS (hemorrhage, increased intracranial pressure, or hypoxic ischemic injury) for other reasons, such as respiratory disease, sepsis, and necrotizing enterocolitis in neonates (NEC). Many different factors, endogenous mediators and mechanisms, and mechanical, can alter vascular pressure. One respiratory condition in pre, near, and at term age infants that results in a composite of neuro-developmental and audiologic impairment (motor, cognitive, perceptual, and behavioral), ranging from between 15-50%, is persistent pulmonary hypertension in the newborn (PPHN) (Lipkin, Davidson, Rhines, & Chang, 2002; Lipkin, Davidson, Rhines, & Chang, 2002). As a respiratory disease process, PPHN can result from pulmonary hypoplasia associated with diaphragmatic, and to a lesser degree abdominal wall hernias, or from vasoconstriction associated with bacterial sepsis, in addition to other pathophysiology (Hagedorn, Gardner, Dickey, & Abman, 2006). This exploratory within group study focuses upon pre, near, and term age infants with differing diagnoses and varying degrees of risk for a diagnoses of CP, developmental coordination disorder, or sensory processing difficulties. Feeding problems are usually prevalent in infants who sustain neurological insult in addition to near term or term age infants with serious developmental disruptions. The investigators measured the intervention effects of neurophysiologically based occupational therapy upon adaptive CNS maturation using several outcome measures. Since infants in the intervention group exhibited a large treatment effect in relationship to their feeding abilities and other covariates, this study should be replicated with infants with similar diagnoses with the same longitudinal outcome measures to learn more about and to further validate the efficacy of neurophysiologically based occupational therapy upon feeding, infant sensorimotor development, and parent efficacy in the NICU.

The following collaborators assisted on this research project:

Walden University: Minneapolis, Minnesota - Ray Thron, PhD, Lela Llorens, Ph.D, OTR, FAOTA, Chester Jones, Ph.D, and Aqueil Ahmad, Ph.D

Primary Children's Medical Center: Salt Lake City, Utah - Mr. Ramsey Worman, Department of Bioengineering, David Bradley, MD and Ms. Barbara Wright, Department of Cardiology, and Mr. Doug Wolfe, Systems Administrator

Mesa State College: Grand Junction, Colorado - Richard Ott, Ph.D, Computer Science, Mathematics, & Statistics

Politecnico di Milano: P.zza Leonardo da Vinci, 32, 20133 Milano, Italy - Manuela Farrario, Ph.D, and Sergio Cerutti, Ph.D. Department of Bioingeneering

ELIGIBILITY:
Inclusion Criteria:

* A mixed group of infants included preterm to term age infants at various levels of risk (per diagnoses) for central nervous system damage and feeding problems; but not small for dates by obstetrical dating and neurological exam, or genetic anomaly. Occupational therapy intervention began per physician approval; when patients were medically stable, and with consistent levels of blood oxygen and stable levels of supplemental oxygen (FiO2), and who were off of medication for paralysis and weaned from sedation. Historical matched control participants were matched with the intervention group participants who have the same diagnosis, gestational age, and neonatal complications.

Exclusion criteria included infants with specific cardiac distress syndrome, genetic anomalies, and small for dates.

Ages: 29 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Null, Jr., M.D., Principal Investigator — University of Utah, Medical Director NCCU, Primary Children's Medical Center; Lynne F. La Corte, Ph.D, OTR/L, OTD, Study Director — University of Utah, Division of Occupational Therapy; Tracy Karp, RNC, MS, NNP, Study Chair — Primary Children's Hospital
Locations (2):
- United States (2):
  - University of Utah / Primary Childrens Medical Center, Salt Lake City, Utah
  - Univesity of Utah / Primary Childrens Medical Center, Salt Lake City, Utah

REFERENCES:
- [Result] La Corte, L.F. (2010). The efficacy of neurophysiologically based occupational therapy intervention in the neonatal intensive care unit: An exploratory study. ProQuest/UMI Dissertation Publishing, no. 3408874. All other citations can be found in the above reference.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 infants were recruited for the study. Later, matched historical controls were utilized for comparison (Nov. 2007-March 2010).
Pre-assignment Details: There were no group assignments. This study was quasi-experimental as matched historical controls were utilized.
Groups:
- Intervention Group: This is the only intervention group that the analysis apply to.
- Matched Historical Comparison Group: Matched Historical Controls drawn from a three year period.
Period: Overall Study
Arm/Group | Intervention Group | Matched Historical Comparison Group
Started | 12 | 10
Completed | 10 | 10
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Matched Historical Comparison Group: This is the only Matched Historical Comparison group infants that the analysis refer to. These infants were drawn from hospital records from a three year period from the time that the study commenced and from the same NCCU. The infants were matched on 19 items modified from Littman and Parmelee (1978) and consisted of four Preterm infants with high risk factors, three term or near term infants with Gastroschisis, two near term infants with Omphalocele, and one near term infant with Congenital Diaphragmatic Hernia.
- Intervention Group: This is the only Matched Historical Comparison group infants that the analysis refer to. The intervention group consisted of four Preterm infants with high risk factors, three term or near term infants with Gastroschisis, two near term infants with Omphalocele, and one near term infant with Congenital Diaphragmatic Hernia.
- Total: Total of all reporting groups
Arm/Group | Matched Historical Comparison Group | Intervention Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: gestational age in weeks] | 34.4 (5.8) | 32.4 (6) | 32.4 (5.8)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: A Priori H1. The Number of Days to Achieve Oral Feeding Between the Intervention Group and the Matched Historical Comparison Group - From All Tube to All Oral Feeding - Was Analyzed.
Description: This outcome measured the number of days it took to go from all tube to all oral feeding or at discharge, whichever came first. Oral feeding percentages were based upon 150 kcal/kg/day. Feeding volumes and weights were taken directly from the nurses notes, and averaged daily. A two sample t-test was used to detect differences between the groups.
Time Frame: The time frame was from Baseline until all oral feeding or discharge, whichever came first (at or before 35 days).
Population: The intervention group and matched historical comparison group consisted of Four pairs of Extremely Preterm to Preterm infants with high risk factors, Three pairs of term or near term infants with Gastroschisis, Two pairs of infants term or near term with Omphalocele, and One pair of infants term age with Congenital Diaphragmatic Hernia.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Intervention Group: This is the only intervention group that the analysis apply to. The intervention and the matched historical comparison group consisted of preterm, near term and full term infants with feeding problems.
- Matched Historical Comparison Group: This is the only Matched Historical Comparison group infants that the analysis refer to. These infants were drawn from hospital records from a three year period from the time that the study commenced and from the same NCCU. The infants were matched on 19 items modified from Littman and Parmelee, (1978).
Arm/Group | Intervention Group | Matched Historical Comparison Group
Number analyzed (Participants) | 10 | 10
Days | 10.8 (5.6) [1.15 to 9.18] | 18.8 (8.2) [1.15 to 9.18]
Statistical Analysis 1: Comparison: Intervention Group vs Matched Historical Comparison Group; The expected outcome was that infants in the intervention group would exhibit significantly less number of days to attain oral feeding; Test type: Superiority or Other; p < 0.005, t-test, 2 sided — The P value is not adjusted for multiple comparisons or for statistical significance; Mean Difference (Net) = 8, 95% CI 2-sided [5 to 11], Standard Error of Mean 1.76

2. Secondary Outcome: A Priori H2: The Increase in Oral Feeding Percentage Over Days Was Correlated With Increasing Respiratory Competency During Oral Feeding; Measured as the High Frequency Percentage (HF%) of Intervention Groups' Heart Rate Variability (HRV) During Feeding.
Description: Oral feeding percentage was based upon 150 kc/kg/day. Heart rate data was recorded about once per week during feeding using a Holter monitor connected to the bedside ecg. This data was downloaded in Cardiology, converted to numerical data as HRV by bioengineers at Politecnico di Milano, Italy. As infants reached 100% of oral feedings, heart rate variability data was analyzed to determine the infants' overall trend toward relaxation, measured as increasing High Frequency Percentage (HF %). Hierarchical linear modeling (HLM) (Singer and Willett, 2003) SPSS Grad Pack 17, mixed model analysis.
Time Frame: The time frame was from Baseline until discharge (at or before 20 days).
Population: The intervention group consisted of Four Preterm infants with high risk factors, Three term or near term infants with Gastroschisis, and Two near term infants with Omphalocele. This outcome measured the correlation between the percentage of oral feedings and the percentage of High Frequesncy Heart Rate Variability.
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- Intervention Group: This is the only intervention group that the analysis apply to and consisted of preterm, near term and full term infants with feeding problems.
Arm/Group | Intervention Group
Number analyzed (Participants) | 9
Percentage
  Percentage of Oral Feeding | 42.60 (33.34) [.99 to 2.79]
  High Frequency Percentage of Heart Rate Var. (HRV) | 34.25 (13.96)
Statistical Analysis 1: Comparison: Intervention Group; Pearson Correlation, 2-tailed; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; This correlation is between the intervention groups' initial level of relaxation and final level of relaxation during the oral feeding period; Slope = 0.275

3. Secondary Outcome: A Priori H3: A Total Score of the Parents' "Global Confidence" (Wolke, 1995) Was Measured on a Pre-post Test Scale.
Description: The Global Confidence Scale of The Mother and Baby Scales (Wolke [in Brazelton and Nugent], 1995]) is a total score measure of mother/parent self efficacy in the NICU as a result of training in NBOTI. It is a total score measure of the parent's perceived efficacy of themselves as confidence in the feeding, handling, caretaking, and interactions needed to foster relationships with their infants. An increase in this score denotes an increase in the parent's perception of their global confidence in caring for their infant. Global Confidence Measure uses a Likert scale. There are three questions, ranging from -3-3. The maximum score is 9, and the minimum score is -9.
Time Frame: Upon an infant's entry into the study, and at discharge (at or less than 20 days).
Population: The intervention group consisted of Three Preterm infants with high risk factors, Three term or near term infants with Gastroschisis, Two near term infants with Omphalocele, and One near term infant Congenital Diaphragmatic Hernia.
Measure: Mean (Standard Deviation); unit: scores on scale
Groups:
- Intervention Group Pre-test: This is the only intervention group that the analysis apply to and consisted of preterm, near term and full term infants with feeding problems.
- Intervention Group Post Test: This is the only intervention group that the analysis apply to.
Arm/Group | Intervention Group Pre-test | Intervention Group Post Test
Number analyzed (Participants) | 9 | 9
scores on scale | 1 (5.9) | 4.56 (4.03)
Statistical Analysis 1: Comparison: Intervention Group Pre-test vs Intervention Group Post Test; Parent pre-post one sided t test of parents' "global confidence", measured parental confidence in feeding, handling, and interacting with their infant; Test type: Superiority or Other; p < .02, t-test, 1 sided; Mean Difference (Net) = 3.6, 95% CI 1-sided [upper limit 6.7], Standard Deviation 5.2 — An increase in this test scale score means more parent confidence

4. Secondary Outcome: A Priori H4: A Total Scale Score of Parents' Perception of "Infant Easiness" (Wolke, 1995) Was Measured on a Pre-post Test Scale.
Description: The Easiness Scale measures the parent's perceived efficacy in the areas of infant irritability, sleeping habits, alertness and responsiveness, and difficulty. The Easiness Scale(Wolke [in Brazelton and Nugent], 1995]) was used to determine mother/parent perceptions of their infants' mood and state in the NICU as a result of training in NBOTI. An increasing score denotes an improvement in parent efficacy in their perception of their infant's easiness.uses a Likert scale. There are four questions, ranging from -3-3. The maximum score is 12, and the minimum score is -12.
Time Frame: Upon an infant's entry into the study, and again at discharge (at or less than 20 days).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on Scale
Arm/Group | Intervention Group Pre-test | Intervention Group Post Test
Number analyzed (Participants) | 9 | 9
Scores on Scale | 3.89 (4.4) | 6.67 (4.03)
Statistical Analysis 1: Comparison: Intervention Group Pre-test vs Intervention Group Post Test; Parent pre-post one sided t test on the Easiness Scale of the Mother and Baby Scales in how parents percieve their interactions (alert-responsiveness, mood) with their infant and infant sleep patterns; Test type: Superiority or Other; p < .03, t-test, 1 sided; Mean Difference (Net) = 2.8, 95% CI 1-sided [upper limit 4.54], Standard Deviation 4.3 — An increase in this test scale score means an increase in the parents' perception of their infants' easiness during caregiving

ADVERSE EVENTS:
Description: Other adverse events were not collected.
Arm/Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The limitation of this study is that the effectiveness of the neurophysiologically based occupational therapy intervention applies to the diagnostic groups of the infants that participated in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No